CLINICAL TRIAL: NCT04641091
Title: Cross-sectional Study of Muscle Perfusion in Patients With PAD by Non-invasive Multispectral Optoacoustic Tomography
Brief Title: Muscle Perfusion in Patients With PAD by Non-invasive MSOT
Status: Completed | Type: Observational
Sponsor: University Hospital Erlangen (Other)
Collaborators: Department of Medicine 1 University Hospital Erlangen, Prof. Dr. Maximilian J. Waldner (Unknown)
Responsible Party: Principal Investigator, Ulrich Rother, PD Dr. med., University Hospital Erlangen
Other Study IDs: MSOT_PAD
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Peripheral Vascular Disease; Peripheral Arterial Disease
Keywords: Peripheral Vascular Disease; Peripheral Arterial Disease; Multispectral Optoacoustic Tomography; Revascularization; Claudicatio intermittens; Critical limb ischemia; MSOT; CLI; PAD; Angiography; Color-Coded Duplex Sonography; CCDS
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group 1: Multispectral Optoacoustic Tomography (MSOT) and B-Mode Ultrasound of the Musculus triceps surae of the affected leg in PAD patients or one leg in healthy volunteers (total 1 site)
  physical assessment: Color-Coded Duplex Sonography / treadmill examination to determine actual walking distance / Ankle-Brachial Index / defined walking distance of 150 meters under medical supervision
  Interventions: Device: Multispectral Optoacustic Tomography (MSOT)
- Study group 2: Multispectral Optoacoustic Tomography (MSOT) and B-Mode Ultrasound of the Musculus triceps surae of the affected leg in PAD patients or one leg in healthy volunteers (total 1 site)
  physical assessment: Color-Coded Duplex Sonography / treadmill examination to determine actual walking distance / Ankle-Brachial Index / defined walking distance of 150 meters under medical supervision
  Interventions: Device: Multispectral Optoacustic Tomography (MSOT)

INTERVENTIONS:
Device: Multispectral Optoacustic Tomography (MSOT) — non-invasive transcutaneous imaging of subcellular muscle components

SUMMARY:
The aim of the proposed study is to define an independent parameter for the diagnostic assessment of the perfusion situation of the calf muscle based on Multispectral Optoacoustic Tomography (MSOT) in a cross-sectional collective of healthy volunteers and patients with PAD. The gold standard is a previously performed angiography of the pelvic and femoral vessels based on routine diagnostics, this Imaging is not mandatory for healthy Control group (study group 1). An independent validation group (study group 2) will validate the results found in study group 1.

DETAILED DESCRIPTION:
Peripheral arterial occlusive disease (PAD) is one of the most common diseases of the elderly with an overall prevalence of about 3-10%. As life expectancy increases, new treatment concepts and new diagnostic procedures are needed. In addition to the possibility of endovascular treatment and open surgery, in some cases there is also the possibility of a conservative therapeutic approach, e.g. with medication.

To date, the only independent non-invasive validation of these treatment options is the measurement of macrocirculation in the form of Color-Coded Vascular Duplex Sonography (CCDS), the Ankle Brachial Index (ABI) or the measurement of walking distance. The S3 guideline for diagnosis, therapy and medical aftercare of PAD published 2015 by the DGA (Deutsche Gesellschaft für Angiologie und Gefäßmedizin [German Society for Angiology and Vascular Medicine]) recommends aftercare in the sense of clinical examinations, especially for patients after vascular surgery. For the validation measures already mentioned, however, there are not infrequent patient groups for which these methods provide only insufficient or unusable results (diabetes mellitus, terminal renal failure). In these cases, independent verification of the success of the therapy performed would have to be performed using angiography (digital subtraction angiography, CT angiography or MR angiography). However, this is not routinely performed in the respective patient populations due to the associated risks (including radiation exposure, contrast agent administration, invasiveness).

Multispectral Optoacoustic Tomography (MSOT) now provides a new non-invasive diagnostic tool that may be able to fill this diagnostic gap.

The aim of this cross-sectional study is to define an independent parameter using the MSOT method, which allows a statement about the current perfusion situation of the lower extremity and correlates with the angiography, which is considered the gold standard. For this purpose, patients of different PAD stages, who already underwent routinely angiographies in advance, will be included. In addition, a control group of healthy volunteers (prior angiography not obligatory) will be examined.

ELIGIBILITY:
Inclusion criteria:

* Patients with manifest PAD stages II - IV according to Fontaine or category 1-6 according to Rutherford
* Adult (>18 years) persons who are able to give their consent
* Patients in whom angiography has been performed as part of routine diagnostics (independent of the study) or in accordance with current guidelines, or has been indicated and the patients has given consent

Exclusion criteria:

* Patients with PAD stage I according to Fontaine or category 0 according to Rutherford
* Underage persons
* Missing consent form
* Patients with manifest PAD in whom angiography is not indicated
* Exclusion due to safety concerns of the study physician (patient with a physical, mental or psychiatric illness which, in the opinion of the study physician, would compromise the safety of the patient or the quality of the data and thus make the patient an unsuitable candidate for the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with
  * PAD IIa with indication for angiography
  * PAD IIb with indication for angiography
  * PAD III with indication for angiography
  * PAD IV with indication for angiography
  who come in for a routine presentation of the vascular surgery consultation hours.
  And healthy volunteers:
  * No PAD previously known
  * No diabetes mellitus previously known
  * No chronic renal insufficiency previously known
  * No symptoms in the sense of a Claudicatio intermitten
  * ABI with normal value
  who are recruted by clinic notices.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Derivation of optimal diagnostic MSOT thresholds for hemoglobin | single time point (1 day)
  Derivation of optimal diagnostic MSOT thresholds for hemoglobin through correlation with TASC classification for angiographic imaging as references for relevant stenosis/ occlusion in patients with PAD

SECONDARY OUTCOMES:
Muscular oxygenated/deoxygenated/total hemoglobin and the MSOT-values at a wavelength of 800nm before and after gait exposure | single time point (1 day)
  Quantitative oxygenated/deoxygenated/total hemoglobin signal and signal at a wavelength of 800 nm (Units: arbitrary units (a. u.)) derived by transcutaneous MSOT in patients with PAD before gait exposure compared to the signals after gait exposure
Correlation of oxygenated/deoxygenated/total hemoglobin content and MSOT-values at a wavelength of 800 nm with the TASC-classification (angiography) | single time point (1 day)
  Quantitative oxygenated/deoxygenated/total hemoglobin signal and signal at a wavelength of 800 nm(Units: arbitrary units (a. u.)) derived by transcutaneous MSOT in patients with PAD correlated with the TASC-classification (angiography)
Difference between oxygenated/deoxygenated hemoglobin before and after gait exposure | single time point (1 day)
  Difference between quantitative oxygenated hemoglobin amount (Units: arbitrary units (a. u.)) and quantitative deoxygenated hemoglobin amount (Units: arbitrary units (a. u.)) derived by transcutaneous MSOT in patients with PAD before gait exposure compared to the amount after gait exposure
Correlation of difference between oxygenated/deoxygenated hemoglobin with the TASC-classification (angiography) | single time point (1 day)
  Difference between quantitative oxygenated hemoglobin amount (Units: arbitrary units (a. u.)) and quantitative deoxygenated hemoglobin amount (Units: arbitrary units (a. u.)) derived by transcutaneous MSOT in patients with PAD correlated with the TASC-classification (angiography)
Muscular quantitative lipid/collagen signal fraction and the MSOT-values at a wavelength of 930 and 1064 nm | single time point (1 day)
  Quantitative lipid/collagen signals and signals at 930 and 1064 nm (Units: arbitrary units (a. u.)) derived by transcutaneous MSOT in patients with different clinical and angiographic PAD stages
Correlation of acquired MSOT parameters with the CCDS flow profile and PSV | single time point (1 day)
  Quantitative oxygenated/deoxygenated/total hemoglobin content and MSOT-values at a wavelength of 800 nm (Units: arbitrary units (a. u.)) derived by transcutaneous MSOT in patients with PAD correlated with the flow profile and PSV of A. CFA and A. poplitea determined by CCDS
Correlation of acquired MSOT parameters with the ABI | single time point (1 day)
  Quantitative oxygenated/deoxygenated/total hemoglobin content and MSOT-values at a wavelength of 800 nm (Units: arbitrary units (a. u.)) derived by transcutaneous MSOT correlated with the ABI
Correlation of acquired MSOT parameters with the walking distance determined by treadmill examination | single time point (1 day)
  Quantitative oxygenated/deoxygenated/total hemoglobin content and MSOT-values at a wavelength of 800 nm (Units: arbitrary units (a. u.)) derived by transcutaneous MSOT correlated with the walking distance determined by treadmill examination
Correlation of acquired MSOT parameters with the clinical severity of PAD | single time point (1 day)
  Quantitative oxygenated/deoxygenated/total hemoglobin content and MSOT-values at a wavelength of 800 nm (Units: arbitrary units (a. u.)) derived by transcutaneous MSOT correlated with the clinical severity of PAD according to Fontaine and Rutherford

CONTACTS AND LOCATIONS:
Locations (1):
- University of Erlangen, Vascular Surgery, Erlangen, Germany

REFERENCES:
- [Background] Lange S, Diehm C, Darius H, Haberl R, Allenberg JR, Pittrow D, Schuster A, von Stritzky B, Tepohl G, Trampisch HJ. High prevalence of peripheral arterial disease and low treatment rates in elderly primary care patients with diabetes. Exp Clin Endocrinol Diabetes. 2004 Nov;112(10):566-73. doi: 10.1055/s-2004-830408. PMID 15578331
- [Background] Alpert JS, Larsen OA, Lassen NA. Exercise and intermittent claudication. Blood flow in the calf muscle during walking studied by the xenon-133 clearance method. Circulation. 1969 Mar;39(3):353-9. doi: 10.1161/01.cir.39.3.353. No abstract available. PMID 4885945

DOCUMENTS (2):
  • Study Protocol (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT04641091/Prot_002.pdf
  • Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT04641091/SAP_003.pdf